CLINICAL TRIAL: NCT07199946
Title: A Phase I/II Double-blind, Randomized, Placebo-controlled Trial to Preserve Residual Insulin Secretion in Children With Recent Onset Type 1 Diabetes by Giving Verapamil
Brief Title: A Phase I/II Trial to Preserve Residual Insulin Secretion in Children With Recent Onset Type 1 Diabetes by Giving Verapamil
Acronym: VERADIAB-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johnny Ludvigsson (Other Government)
Collaborators: Region Östergötland (Other); Region Jönköping County (Other Government)
Responsible Party: Sponsor-Investigator, Johnny Ludvigsson, Professor, Linkoeping University
Organization: Linkoeping University (Other Government)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202100-3096; 2024-515106-30-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-26; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes
Keywords: c-peptide; beta cell function; children; Verapamil
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Verapamil

STUDY DESIGN:
Intervention Model Description: Part A open study including 6 patients, and thereafter part B, a double-blind, randomized, placebo-controlled trial including 30 patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part A: Open label intervention for 6 patients (Experimental): Intervention: Open label pilot arm with Verapamil treatment
  Interventions: Drug: Verapamil (Part A)
- Part B: Active treatment with Verapamil in a double blind randomized controlled trial (Active Comparator): Active treatment with Verapamil 3-6 mg/ kg body weight and 24 hrs in a double blind randomized controlled trial
  Interventions: Drug: Verapamil (Part A)
- Part B: Placebo arm in a double blind randomized controlled trial (Placebo Comparator): Placebo given in the same way and times as the active treatment, for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Verapamil (Part A) — Verapamil 3-6mg/kg body weight and 24 hrs
  Other Names: Isoptin
  Arms: Part A: Open label intervention for 6 patients; Part B: Active treatment with Verapamil in a double blind randomized controlled trial
Drug: Placebo — Placebo given in part B, the comparator arm of the double blind randomized trial
  Arms: Part B: Placebo arm in a double blind randomized controlled trial

SUMMARY:
The objective of this trial is first to evaluate safety and then the effect on preservation of residual beta cell function also clinical efficacy by treatment with Verapamil in children with recent onset Type 1 diabetes.

Patients are included with the following inclusion criteria;

* Informed consent given by patients and caregivers/parents Type 1 diabetes according to the ADA classification within the previous 3 months at the time of screening
* Age 4.00 -9.99 years at Diagnosis of Type 1 diabetes
* Fasting C-peptide >0.12 nmol/ml
* Elevated levels of any diabetes-related antibody/ies (eg GADA, IAA, IA-2A, ZnT8A ) is/are present.

While they are not allowed to participate if they eg have previous cardiac problems or abnormal ECG.

The study is a Phase I/II trial, with two parts: A. 6 patients participate in an open controlled study without any placebo with the primary aim to evaluate safety. After a baseline evaluation including ECG, physical examination, mixed Meal Tolerance Test evaluating residual beta cell fuction, these patients will be treated for 12 months with Verapamil 3-6 mg/kg body weight/24 hrs, divided into two daily doses. When these 6 patients have been followed for 6 months, and safety and tolerability is regarded as good, part B will start: In part B the next 30 patients will be randomized 1:1 in a double-blind placebo-controlled study into two arms: 15 patients will receive active treatment for 12 months with Verapamil 3-6 mg/kg body weight/24 hrs divided into two daily oral doses, while 15 patients will receive placebo in two daily doses for 12 months. Efficacy will be evaluated with MMTT and clinical response ( insulin dose/kg body weight/24 hrs, HbA1c, and CGM data on Glucose Time in Range), from baseline and after 12 and 24 months.

There is a great benefit of preservation of residual insulin secretion, and therefore therapies aiming at preservation of this function justifies treatments that are quite heavy, even dangerous and expensive.

In this study the investigators will use oral Verapamil, a drug which is used as antihypertensive treatment in different ages, even in children in the neonatal period, with limited adverse events and risks. Verapamil treatment has shown encouraging results preserving beta cell function in Type 1 diabetes in adults, and the investigators expect to get similar positive effects also in young children, in whom so far no immune intervention has shown efficacy.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is by far the most common chronic, serious, life-threatening disease in Sweden, and tends to become an extremely serious global problem. Residual insulin secretion is of crucial importance to facilitate treatment, prevent acute and late complications and improve quality of life.

Primary objective: To evaluate the effect on preservation of residual beta cell function but treatment with Verapamil Secondary objectives: To evaluate safety, but also clinical efficacy of Verapamil treatment such as blood glucose control and prevention of acute complications, and immunological effect on the disease process

Primary outcome:

• Change in C-peptide AUCmean 0-120 min) during an MMTT from baseline to month 24.

Secondary outcome:

* Change in C-peptide fasting and 90 minute value during an MMTT from baseline to month 24
* Proportion of patients with peak C-peptide > 0.20 nmol/l at month 24
* Hemoglobin A1c (HbA1c), change between baseline and subsequent visits
* Exogenous insulin dose per kg body weight and 24 hours, change between baseline and subsequent visits
* Safety and tolerability

Trial population:

Patients must be 4.0 - 9.99 years old, and diagnosed with type 1 diabetes (T1D) within the previous 3 months at the time of screening.

Number of subjects: Part A: 6 Part B: 30 (In total 36)

Inclusion criteria:

* Informed consent given by patients and caregivers/parents Type 1 diabetes according to the ADA classification within the previous 3 months at the time of screening
* Age 4.00 -9.99 years at Diagnosis of Type 1 diabetes
* Fasting C-peptide >0.12 nmol/ml
* Elevated levels of any diabetes-related antibody/ies (eg GADA, IAA, IA-2A, ZnT8A ) is/are present.

Exclusion criteria:

* Cardiac disease/ problems
* Abnormal ECG
* history of abnormal blood pressure
* Previous or current treatment with immunosuppressant therapy (although topical or inhaled steroids are accepted)
* Continuous treatment with any inflammatory drug (sporadic treatment e.g. because of headache or in connection with fever a few days will be accepted)
* Treatment with any oral or injected anti-diabetic medications other than insulin
* A history of anaemia or significantly abnormal haematology results at screening
* Participation in other clinical trials with a new chemical entity within the previous 3 months
* Inability or unwillingness to comply with the provisions of this protocol
* A significant illness other than diabetes within 2 weeks prior to first dosing. However treated celiac disease and hypothyroidism with adequate treatment will be accepted.
* Deemed by the investigator not being able to follow instructions and/or follow the study protocol

Intervention:

The study is a Phase I/II trial, with two parts: A. 6 patients participate in an open controlled study without any placebo with the primary aim to evaluate safety. After a baseline evaluation including ECG, physical examination, mixed Meal Tolerance Test evaluating residual beta cell fuction, these patients will be treated for 12 months with Verapamil 3-6 mg/kg body weight/24 hrs, divided into two daily doses. When these 6 patients have been followed for 6 months, and safety and tolerability is regarded as good, part B will start: In part B the next 30 patients will be randomized 1:1 in a double-blind placebo-controlled study into two arms: 15 patients will receive active treatment for 12 months with Verapamil 3-6 mg/kg body weight/24 hrs divided into two daily oral doses, while 15 patients will receive placebo in two daily doses for 12 months. Efficacy will be evaluated with MMTT and clinical response ( insulin dose/kg body weight/24 hrs, HbA1c, and CGM data on Glucose Time in Range), from baseline and after 12 and 24 months.

Investigational medicinal product(s), dosage, administration: 3-6 mg/kg body weight/24 hrs of Verapamil ( Isoptin) is given per os two times per day Ethical considerations, benefit/risk: There is a great benefit of preservation of residual insulin secretion, and therefore therapies aiming at preservation of this function justifies treatments that are quite heavy, even dangerous and expensive. Thus it has been regarded as justified to treat even children with Type 1 diabetes at onset with drugs like monoclonal antibodies against the CD3-receptor, which causes adverse events in principally all patients, some even quite serious adverse events and risks. Even cytostatics have been used.

The investigators will here use oral Verapamil, a drug which is used as antihypertensive treatment in different ages, even in children in the neonatal period, with limited adverse events and risks. Verapamil treatment has shown encouraging results preserving beta cell function in Type 1 diabetes in adults, and the investigators expect to get similar positive effects also in young children, in whom so far no immune intervention has shown efficacy.

Thus, there is a clear possibility of therapeutic benefit, whereas the risk is very small, which makes the trial ethically justified.

ELIGIBILITY:
Inclusion criteria: • Informed consent given by patients and caregivers/parents

* Type 1 diabetes according to the ADA classification within the previous 3 months at the time of screening
* Age 4.00 -9.99 years at Diagnosis of Type 1 diabetes
* Fasting C-peptide >0.12 nmol/ml
* Elevated levels of any diabetes-related antibody/ies (eg GADA, IAA, IA-2A, ZnT8A ) is/are present.

Exclusion criteria: • Cardiac disease/problems, abnormal ECG, or history of abnormal blood pressure

* Previous or current treatment with immunosuppressant therapy (although topical or inhaled steroids are accepted)
* Continuous treatment with any inflammatory drug (sporadic treatment e.g. because of headache or in connection with fever a few days will be accepted)
* Treatment with any oral or injected anti-diabetic medications other than insulin
* A history of anaemia or significantly abnormal haematology results at screening
* Participation in other clinical trials with a new chemical entity within the previous 3 months
* Inability or unwillingness to comply with the provisions of this protocol
* A significant illness other than diabetes within 2 weeks prior to first dosing. However treated celiac disease and hypothyroidism with adequate treatment will be accepted.
* Deemed by the investigator not being able to follow instructions and/or follow the study protocol

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Change in C-peptide AUCmean 0-120 min) during an MMTT from baseline to month 24. | 24 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0". | 24 months
  Adverse events are registered after history, clinical examinations, laboratory tests and ECG. Patients and parents are interviewed about tolerability

SECONDARY OUTCOMES:
Change in C-peptide fasting and 90 minute value during an MMTT from baseline to month 24 | 24 months
Proportion of patients with peak C-peptide > 0.20 nmol/l at month 24 | 24 months
Hemoglobin A1c (HbA1c), change between baseline and subsequent visits | 24 months
Insulin dose/kg body weight/24 hrs | 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Pediatric Clinic , Ryhovs hospital, Jönköping
  - Crown Princess Victoria Children´s Hospital, University Hospital, Linköping